CLINICAL TRIAL: NCT02308891
Title: Multicenter Prospective Randomized Trial of Aggressive Hydration Strategy to Reduce Post-ERCP Pancreatitis
Brief Title: A Prospective Trial of Aggressive Hydration Strategy to Reduce Post-ERCP Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dankook University (Other)
Collaborators: Wonkwang University (Other); University of Ulsan (Other)
Responsible Party: Principal Investigator, Jun Ho Choi, Assistant Professor, Dankook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2014-09-011
Record Dates: First submitted 2014-11-26; First posted 2014-12-04 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Post-ERCP Acute Pancreatitis
Keywords: pancreatitis; ERCP
MeSH Terms: conditions — Pancreatitis | interventions — Ringer's Lactate; Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vigorous hydration arm (Experimental): Patients will be randomly allocated to vigorous hydration arm. Patients in the vigorous hydration arm will receive fluids via infusion by the following protocol.
  * Initial bolus of lactated Ringer's solution at 10mL/kg over 1 hour prior to ERCP
  * Intravenous lactated Ringer's solution at a rate of 3mL/kg/h during the procedure and continued for 8 hours.
  * At the end of ERCP, post-procedure bolus of lactated Ringer's solution at 10mL/Kg over 1hour
  Interventions: Drug: lactated Ringer's solution (vigorous hydration arm); Device: endoscopic retrograde cholangiopancreatography (ERCP)
- standard hydration arm (Active Comparator): Patients will be randomly allocated to standard hydration arm. Patients in the standard hydration arm will receive fluids via infusion by the following protocol.
  - Patients will receive lactated Ringer's solution at the start of the ERCP and the fluids will be administered at a rate of 1.5ml/kg/h during the procedure and for 8hours after ERCP.
  Interventions: Drug: lactated Ringer's solution (standard hydration arm); Device: endoscopic retrograde cholangiopancreatography (ERCP)

INTERVENTIONS:
Drug: lactated Ringer's solution (vigorous hydration arm) — * Initial bolus of lactated Ringer's solution at 10mL/kg over 1 hour prior to ERCP
  * Intravenous lactated Ringer's solution at a rate of 3mL/kg/h during the procedure and continued for 8 hours.
  * At the end of ERCP, post-procedure bolus of lactated Ringer's solution at 10mL/Kg over 1hour
  Arms: vigorous hydration arm
Drug: lactated Ringer's solution (standard hydration arm) — - Patients will receive lactated Ringer's solution at the start of the ERCP and the fluids will be administered at a rate of 1.5ml/kg/h during the procedure and for 8hours after ERCP.
  Arms: standard hydration arm
Device: endoscopic retrograde cholangiopancreatography (ERCP) — endoscopic retrograde cholangiopancreatography

SUMMARY:
Postendoscopic retrograde cholangiopancreatography pancreatitis is the most frequent and serious complication of ERCP procedures, occurring in approximately 5-15% of unselected patients. Pharmacologic prevention of post-ERCP pancreatitis has been the topic of several investigations in recent years. Hydration is considered a mainstay of treatment for acute pancreatitis. We perform multicenter, prospective, randomized trial to investigate whether intravenous vigorous hydration with lactated Ringer's solution reduces the risk of post-ERCP pancreatitis.

Inclusion criteria : consecutive patients older than 18 years who are scheduled to undergo diagnostic or therapeutic ERCP will be recruited.

Patients will be randomly assigned in a 1:1 ratio to receive either vigorous hydration (treatment arm) or standard hydration (standard arm). Randomization will be performed in a double blinded fashion using computer-generated random numbers.

Treatment arm (vigorous hydration arm);

* Initial bolus of lactated Ringer's solution at 10 mL/kg over 1 hour prior to ERCP
* Intravenous lactated Ringer's solution at a rate of 3 mL/kg/h during the procedure and continued for 8 hours.
* At the end of ERCP, post-procedure bolus of lactated Ringer's solution at 10 mL/Kg over 1hour Standard arm (standard hydration arm);
* Patients will receive lactated Ringer's solution at the start of the ERCP and the fluids will be administered at a rate of 1.5 ml/kg/h during the procedure and for 8hours after ERCP.

The primary endpoint was development of post-ERCP pancreatitis, which define as increased pancreatic pain (more than 3 on a visual analogue pain scale) and hyperamylasemia (three times the upper limit of normal).

The secondary endpoint included the development of asymptomatic hyperamylasemia, severity of pancreatitis, and fluid overload.

DETAILED DESCRIPTION:
Postendoscopic retrograde cholangiopancreatography pancreatitis is the most frequent and serious complication of ERCP procedures, occurring in approximately 5-15% of unselected patients. Pharmacologic prevention of post-ERCP pancreatitis has been the topic of several investigations in recent years. Hydration is considered a mainstay of treatment for acute pancreatitis. We perform multicenter, prospective, randomized trial to investigate whether intravenous vigorous hydration with lactated Ringer's solution reduces the risk of post-ERCP pancreatitis.

Patients will be randomly assigned in a 1:1 ratio to receive either vigorous hydration (treatment arm) or standard hydration (standard arm). Randomization will be performed in a double blinded fashion using computer-generated random numbers.

Treatment arm (vigorous hydration arm);

* Initial bolus of lactated Ringer's solution at 10 mL/kg over 1 hour prior to ERCP
* Intravenous lactated Ringer's solution at a rate of 3 mL/kg/h during the procedure and continued for 8 hours.
* At the end of ERCP, post-procedure bolus of lactated Ringer's solution at 10 mL/Kg over 1 hour

Standard arm (standard hydration arm);

- Patients will receive lactated Ringer's solution at the start of the ERCP and the fluids will be administered at a rate of 1.5 ml/kg/h during the procedure and for 8hours after ERCP.

The primary endpoint is development of post-ERCP pancreatitis, which define as increased pancreatic pain (more than 3 on a visual analogue pain scale) and hyperamylasemia (three times the upper limit of normal).

The secondary endpoint included the development of asymptomatic hyperamylasemia, severity of pancreatitis, and fluid overload.

Serum amylase levels are measured at baseline, and at 8 hours and 18-24 hours, 48 hours after the procedure.

Investigators recorded the details of the maneuvers performed, including:

1. the total time of the procedure,
2. the number of attempts at cannulation,
3. the number of pancreatic duct cannulation,
4. the final diagnosis by ERCP,
5. whether a sphincterotomy, a needle-knife papillotomy, or stent placement
6. endoscopic papillary balloon dilation,
7. common bile duct (C) tissue sampling (biopsy, brush, cytology),
8. common bile duct-intraductal ultrasonography (C-IDUS),

   * Serum amylase is determined 8, 18~24, and 48 hours after ERCP.

     * If the 12-hours serum amylase level was > 3 times the upper normal limit and the patient exhibited pain or nausea and vomiting, then the patient had pancreatitis.
     * Acute pancreatitis is defined as serum amylase > 3 times the upper limit of normal and associated with epigastric pain, back pain, and epigastric tenderness.
   * Statistical analysis:

     1. Randomization was done by the GI nurse, concealed envelop
     2. Data were summarized by descriptive statistics.
     3. The Chi square was used to compare categorical patient data.
     4. The Student's t test was used to compare continuous variables.
     5. Two-tailed P < 0.05 was considered to indicate significance.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients older than 18 years who are scheduled to undergo diagnostic or therapeutic ERCP will be recruited

Exclusion Criteria:

* Patients will be excluded if they have acute pancreatitis during the 2 weeks before ERCP, a history of chronic pancreatitis, previous sphincterotomy, or if they refuse to participate the study protocol. Patients will be also excluded if they undergo ERCP, for procedures such as stone removal following previous sphincterotomy, change or removal of previous biliary stents, or surveillance biopsy after endoscopic papillectomy without pancreatography, which are considered to carry minimal risks of post-ERCP pancreatitis. Patients with high risk of fluid overload (heart failure, more than NYHA II; renal insufficiency, creatinine clearance <40ml/min; liver cirrhosis; or hypoxemia, SaO2 <90%; signs of pulmonary edema) are excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
development of post-ERCP pancreatitis | 48 hours
  define as increased pancreatic pain (more than 3 on a visual analogue pain scale) and hyperamylasemia (three times the upper limit of normal).

SECONDARY OUTCOMES:
development of hyperamylasemia | 48 hours
  hyperamylasemia (three times the upper limit of normal).
severity of pancreatitis | 3 months
  pancreatitis criteria
any signs of fluid overload | 48 hours
  pulmonary or peripheral edema

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ho Choi, MD, Principal Investigator — Dankook University College of Medicine
Locations (3):
- South Korea (3):
  - Dankook University College of Medicine, Cheonan, Chungcheongnam-do
  - Wonkwang University, Iksan, Jeollabukdo
  - University of Ulsan, Ulsa University Hospital, Ulsan

REFERENCES:
- [Derived] Choi JH, Kim HJ, Lee BU, Kim TH, Song IH. Vigorous Periprocedural Hydration With Lactated Ringer's Solution Reduces the Risk of Pancreatitis After Retrograde Cholangiopancreatography in Hospitalized Patients. Clin Gastroenterol Hepatol. 2017 Jan;15(1):86-92.e1. doi: 10.1016/j.cgh.2016.06.007. Epub 2016 Jun 14. PMID 27311618